CLINICAL TRIAL: NCT05645900
Title: Immunogenicity and Safety of a Quadrivalent Influenza Virus Subunit Vaccine in Subjects Aged 6-35 Months : A Randomized, Double-blind, Active-controlled Phase III Trial
Brief Title: A Clinical Trial of an Quadrivalent Influenza Virus Subunit Vaccine in Chinese Children Aged 6 to 35 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ab&B Bio-tech Co., Ltd.JS (Other)
Collaborators: Henan Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017L04970/1-3
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental vaccine 1 (Experimental): Subjects received 2 doses of 0.5 mL of quadrivalent influenza virus subunit vaccine, 28 days apart
  Interventions: Biological: Quadrivalent influenza virus subunit vaccine
- experimental vaccine 2 (Experimental): Subjects received 2 doses of 0.25 mL of quadrivalent influenza virus subunit vaccine, 28 days apart
  Interventions: Biological: Quadrivalent influenza virus subunit vaccine
- control vaccine (Active Comparator): Subjects received 2 doses of 0.25 mL of Quadrivalent split influenza virus vaccine, 28 days apart
  Interventions: Biological: Quadrivalent split influenza virus vaccine

INTERVENTIONS:
Biological: Quadrivalent influenza virus subunit vaccine — This vaccine（0.5ml） is produced by Ab&b Biotechnology Co., Ltd.JS。Subjects will receive two doses of quadrivalent influenza virus subunit vaccine administered 28 days apart by intramuscular injection
  Arms: experimental vaccine 1
Biological: Quadrivalent influenza virus subunit vaccine — This vaccine（0.25ml） is produced by Ab&b Biotechnology Co., Ltd.JS。Subjects will receive two doses of quadrivalent influenza virus subunit vaccine administered 28 days apart by intramuscular injection
  Arms: experimental vaccine 2
Biological: Quadrivalent split influenza virus vaccine — This vaccine（0.25ml） is produced by HUALAN BIO。Subjects will receive two doses of quadrivalent split influenza virus vaccine administered 28 days apart by intramuscular injection
  Arms: control vaccine

SUMMARY:
A random, blind and positive control design was adopted.the investigators will assess the safety and immunogenicity of 2 doses of an quadrivalent influenza vaccine virus subunit in children aged 6 to 35 months.

A total of 2,772 subjects in the 6-35 month age group were randomly divided into experimental vaccine 1, experimental vaccine 2 and control vaccine groups at a ratio of 1:1:1, and received the corresponding vaccine respectively. 2 doses in the whole course, 28 days apart.

Safety observation: All subjects received 30 minutes of immediate response observation after each dose of vaccine and 0-7 days of systematic active safety observation; After 7 days of vaccination, the incidence of adverse events was observed by combining regular weekly follow-up with subject's voluntary report. Safety observation was conducted for 0-28/30 days after each dose of vaccine. Serious adverse events (SAE) were collected within 6 months after the first dose was administered.

Immunogenicity observation: Blood samples were collected before the first dose and 28 days after the full dose for influenza virus HI antibody detection.

Observation of immune persistence: Blood samples of 3 and 6 months after immunity were collected for influenza virus HI antibody detection.

ELIGIBILITY:
Inclusion Criteria:

* 6-35 months healthy infants;
* The legal guardian voluntarily consented to the subject's participation in the study, and the legal guardian/trustee signed the Informed Consent Form and complied with the requirements of the protocol.

Exclusion Criteria:

1. Exclusion criteria for the first dose:

   * Armpit temperature ≥37.3℃ on the day of enrollment;
   * Persons infected with influenza virus confirmed by laboratory testing within the previous 6 months;
   * Received any influenza vaccine (registered or experimental) within the previous 12 months or planned to receive any influenza vaccine during the study period;
   * Allergic to any components of the vaccine, such as eggs, excipients, formaldehyde, etc;
   * Previous history of severe allergy to any vaccine or drug (e.g., but not limited to: anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local anaphylactic necrosis reaction (Arthus reaction);
   * 6-23 months: premature (delivered before the 37th week of gestation), low weight (birth weight <2500g) , or a history of dystocia, asphyxia rescue, and neurological damage;
   * Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc;
   * Acute disease, serious chronic disease or acute attack of chronic disease on the day of vaccination;
   * Congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), juvenile rheumatoid arthritis (JRA), or other autoimmune diseases;
   * History of asthma, instability within the past two years requiring emergency treatment, hospitalization, intubation, oral or intravenous corticosteroids;
   * Progressive neurological disease, history of seizures, epilepsy, encephalopathy, Guillain-Barre syndrome, or history or family history of mental illness;
   * Suffering from serious cardiovascular disease (heart disease, pulmonary heart disease, pulmonary edema);
   * Asplenia, functional asplenia, and asplenia or splenectomy resulting from any condition; Resection or partial resection of other important organs;
   * History of coagulation dysfunction (e.g., coagulation factor deficiency, coagulation disease);
   * A history of live attenuated vaccine vaccination within 14 days and a history of other vaccines within 7 days before vaccination;
   * Immune-boosting or suppressant therapy within 3 months (continuous oral or intravenous infusion for more than 14 days);
   * Received blood or blood-related products;
   * Plan to relocate prior to the completion of the study or to be away for an extended period during the scheduled study visit;
   * Being or planning to participate in other clinical trials in the near future;
   * Any ineligibility to participate in the trial was determined by the investigator.
2. Exclusion criteria for the second dose:

   * Severe allergic reaction after the first dose of vaccine;
   * Serious adverse reactions related to the first dose of vaccine;
   * The investigator will decide whether to continue to participate in the study if new findings or new occurrence after the first dose inoculation do not meet the inclusion criteria of the first dose or the exclusion criteria of the first dose;
   * Other reasons for exclusion, according to the investigator.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2772 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events/reactions within 30 minutes after each dose of inoculation | Within 30 minutes after each dose
  Occurrence of adverse events/reactions within 30 minutes after each dose of inoculation
Occurrence of adverse events/reactions within 0-7 days after each dose of inoculation | Within 0-7 days after each dose
  Occurrence of adverse events/reactions within 0-7 days after each dose of inoculation
Occurrence of adverse events/reactions within 8-28/30 days after each dose of inoculation | Within 8-28/30 days after each dose
  Occurrence of adverse events/reactions within 8-28/30 days after each dose of inoculation
Occurrence of serious adverse events within 6 months from the first dose to the full course of vaccination | Within 6 months from the first dose to the full course of vaccination
  Occurrence of serious adverse events within 6 months from the first dose to the full course of vaccination
The seroconversion rates ,the proportion of antibody titer ≥1:40, and the GMT at 28 days after full immunization | At 28 days after full immunization
  The seroconversion rates ,the proportion of antibody titer ≥1:40, and the GMT at 28 days after full immunization

SECONDARY OUTCOMES:
The seroconversion rates ,the proportion of antibody titer ≥1:40, and the GMT at 3 months after full immunization | At 3 months after full immunization
  The seroconversion rates ,the proportion of antibody titer ≥1:40, and the GMT at 3 months after full immunization
The seroconversion rates ,the proportion of antibody titer≥1:40, and the GMT 6 months after full immunization | At 6 months after full immunization
  The seroconversion rates ,the proportion of antibody titer≥1:40, and the GMT 6 months after full immunization

CONTACTS AND LOCATIONS:
Locations (1):
- Ab&b Biotechnology Co., Ltd.JS, Taizhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No